CLINICAL TRIAL: NCT00330954
Title: Gene Expression Profiling in Type 1 Diabetes
Status: Completed | Type: Observational
Sponsor: Children's Mercy Hospital Kansas City (Other)
Responsible Party: Karen Kover, PhD, Children's Mercy Hospitals and Clinics
Other Study IDs: 06 05-087E
Record Dates: First submitted 2006-05-26; First posted 2006-05-29 (Estimated); Last update posted 2010-03-05 (Estimated); Status verified 2010-03

CONDITIONS: Type 1 Diabetes Mellitus
Keywords: viral response genes
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole Blood saved frozen for 1 year
Oversight: Data Monitoring Committee: No

SUMMARY:
One of the goals of the Kansas City Diabetes Consortium is to identify and characterize genes and their products that are associated with T1DM. Characterization of such genes and their products can aid in developing new tools for risk assessment, development of new prevention strategies and monitoring progression of disease.

Study design: Descriptive, basic science pilot study. The results of this pilot study will be used to help design a much larger study to address the importance of viral response and autoimmune diabetes.

DETAILED DESCRIPTION:
The hypothesis is that viral responsive genes are up-regulated prior to the onset of symptoms of Type 1 Diabetes (T1DM) and may correlate with increased expression of interferon alpha.

Both genetic and environmental factors contribute to risk of development of T1DM. There are a number of conflicting reports associating viral infections and T1DM in genetically susceptible individuals and causality has not been proven. Viruses may not have a large role in the initiation of islet cell autoimmunity but more of a role in acceleration of the disease leading to overt symptoms. There are no studies describing viral responsive gene expression in these individuals.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects 7-14 years of age
* New onset T1DM
* Five years post onset of T1DM
* Participant in the TrialNet initiative and either antibody positive or antibody negative sibling control
* Body weight sufficient to tolerate an additional 15ml (1 tbsp) blood loss

Exclusion Criteria:

* Subjects who do not meet the criteria above
* Subjects who have received steroids or other immunosuppressive therapy within the 6 months prior to enrollment into the study

Ages: 7 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Male and female subjects 7-14 years of age
  * New onset T1DM
  * Five years post onset of T1DM
Sampling Method: Non-Probability Sample
Enrollment: 64 (Estimated)
Dates: Start 2006-06; Study Completion 2008-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Karen Kover, PhD, Principal Investigator — Children's Mercy Hospital Kansas City
Locations (1):
- Children's Mercy Hospital, Kansas City, Missouri, United States